CLINICAL TRIAL: NCT03033940
Title: Kinematics Analysis: Comparison Between the Cruciate Retaining, Fixed Bearing Primary Total Knee Arthroplasty ATTUNE TM Knee System and the Fixed Bearing PFC Sigma Curved Total Knee Arthroplasty
Brief Title: Total Knee Arthroplasty Videofluoroscopy
Status: Completed | Type: Observational
Sponsor: Dr. Renate List (Other)
Responsible Party: Sponsor-Investigator, Dr. Renate List, Dr. sc. ETH, Group Leader Clinical Movement Biomechanics, Senior Research Associate, Institute for Biomechanics, ETH Zürich
Organization: Institute for Biomechanics, ETH Zürich (Other)
Other Study IDs: ATTUNE-SIGMA-2016
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Total Knee Anthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ATTUNE TM subjects
  Interventions: Radiation: Observational use of fluoroscopy
- PFC Sigma subjects
  Interventions: Radiation: Observational use of fluoroscopy

INTERVENTIONS:
Radiation: Observational use of fluoroscopy

SUMMARY:
The primary objective is to quantify and compare the three-dimensional kinematics of the cruciate retaining (CR), fixed bearing ATTUNETM TKA to the kinematics of the PFC Sigma Curved CR Fixed Bearing TKA (both DePuy Synthes, Johnson and Johnson) during daily activities.

The secondary objective is to describe the kinematics in terms of range of motion, patterns of anterior-posterior motion of the nearest medial and lateral points ("posterior femoral rollback") and tibio-femoral internal/external rotation as well as the kinetics during daily activities, such as level gait, a deep knee bend (only ATTUNETM subjects), sitting down onto a chair, standing up from a chair and stair descent by means of video-fluoroscopy.

Furthermore, the encoded data will be handed over to DePuy Synthes (Johnson and Johnson) and to the Center for Orthopaedic Engineering of the University of Denver, where it will be used within a musculoskeletal model with the aim of simulating tibiofemoral contact mechanics and changes in the musculoskeletal system due to the TKA.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral TKA (ATTUNETM/Sigma) due to osteoarthritis
* BMI ≤ 33
* Good clinical outcome, KOOS > 70
* No or very low pain VAS < 2
* At least one year post-op
* Standardized general health survey score (SF-12) within the normal range for people in their age group

Exclusion Criteria:

* Actual significant problem on lower extremities
* Misaligned TKA
* Any other arthroplasty at the lower extremities
* Patient incapable to understand and sign informed consent
* Incapable of performing the motion tasks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational study on 15 subjects with the ATTUNE TM CR Fixed Bearing TKA and 15 subjects with PFC Sigma Curved CR Fixed Bearing TKA during level walking, deep knee bend (only ATTUNE TM subjects), sitting down onto a chair, standing up from a chair and stair descent. The present study extends the subject groups of a previous feasibility study (KEK-ZH-Nr. 2014-0468) from 5 to 15 ATTUNE TM and from 6 to 15 PFC Sigma Curved CR Fixed Bearing TKA subjects. Based on a power analysis of the existing data of 5 ATTUNE TM subjects and 6 subjects with a PFC Sigma Curved CR Fixed Bearing TKA in the previous feasibility study (KEK-ZH-Nr. 2014-0468) the minimal sample size for the comparative evaluation of 15 subjects within each group was estimated. The participants must be able to perform the daily activity tasks mentioned above
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the three-dimensional kinematics of the cruciate retaining (CR), fixed bearing ATTUNETM TKA to the kinematics of the PFC Sigma Curved CR Fixed Bearing TKA | 3 hours
  With video-fluoroscopic assessment it is possible to directly measure the kinematics of the tibial and the femoral components in vivo during daily activities, such as level walking, a deep knee bend (only ATTUNETM subjects), sitting down onto a chair, standing up from a chair and stair descent. Thus, for the first time the present study provides in vivo assessed data of the 3D motion of the ATTUNETM System during daily activities and allows a comparison to a conventional TKA based on the same methodology. The knowledge of the in vivo kinematic behaviour of the ATTUNETM System in comparison to the conventional TKA leads to an improved understanding of the design principle.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Biomechanics, ETH Zurich, Zurich, Switzerland